CLINICAL TRIAL: NCT02168959
Title: Postoperative Pain Management With a Continuous Femoral Nerve Block in Patients With a Tibial Plateau Fracture
Brief Title: Continuous Femoral Nerve Block With a Tibial Plateau Fracture
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Eric Kubiak, M.D., University of Utah
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 56481
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Tibial Plateau Fracture
Keywords: Femoral Nerve Block; Pain Control; Tibial Plateau Fracture; Prospective; Randomized
MeSH Terms: conditions — Tibial Plateau Fractures; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Femoral nerve block (Active Comparator): bupivacaine
  Interventions: Drug: bupivacaine
- No femoral nerve block (No Intervention): No block

INTERVENTIONS:
Drug: bupivacaine — This drug is standard of care. The point of the study is to see if this method will yield better pain scores and improved patient satisfaction vs. non-nerve block. Simply: prospective observation of two standard methods.
  Arms: Femoral nerve block

SUMMARY:
The primary purpose of the proposed study is to compare postoperative pain scores and total opioid consumption between two groups randomized to either receive or not receive a femoral nerve block for pain control following surgical repair of a tibial plateau fracture. Pain will be assessed post-operatively using standard numeric pain scores rated on a 0 - 10 scale, as well as using the University new pain assessment tool - the Clinically Aligned Pain Assessment (CAPA). This new 5 question pain assessment tool has not yet been validated, but does address several key questions, including patient comfort, pain control, change in pain status, daily functioning, and sleep quality. Along with post-operative pain scores, we will compare total opioid consumption between the two groups.

The null hypothesis is that there is no difference in pain scores or total opioid consumption between patients receiving a femoral nerve block and those without a nerve block following surgical repair of a tibial plateau fracture.

A secondary outcome will examine long-term pain control, range of motion, and functional status of these patients at their regular orthopedic clinic follow-up appointments. The same pain scores will be assessed, along with quadriceps strength and knee range of motion. Patients will complete the PROMIS Physical Function CAT and short Musculoskeletal Function Assessment, patient reported outcomes tools to evalute physical function.

A teriary outcome will be to retrospectively examine postoperative pain scores and total opioid consumption for all tibial plateau fracture patients seen at the University of Utah for surgical repair in the past 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, aged 18 years or older, who are presenting to the University Hospital for surgical repair of a tibial plateau fracture will be considered for inclusion in the prospective study. The diagnosis of a tibial plateau fracture and the decision to proceed to the operating room for surgery will be made by the attending surgeon of the orthopedic trauma service based on his expertise and standard of care.
* Male and female patients, aged 18 years or older, who have underwent surgery performed by Dr. Kubiak or Dr. Higgins at University Hospital for repair of a tibial plateau fracture will be considered for inclusion in the retrospective study.

Exclusion Criteria:

Prospective Study:

* Patients who do not speak English
* Patients who are unable to effectively communicate with their treatment team (example: mechanically ventilated patients and mentally handicapped patients)
* Patients less than 18 years old
* Patients with ongoing compartment syndrome
* Patients with an allergy or intolerance to bupivacaine
* Patients with other significant associated traumatic injuries that would be expected to delay their overall recovery (example: a patient who sustains a motor vehicle accident and fractures their tibia but also sustains massive intra-abdominal injury with serious damage to their liver and other vital organs)
* Patients with ipsilateral femoral fractures

Retrospective:

* Patients less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Score and patient satisfaction | Follow-up Visits up to 1-Year

SECONDARY OUTCOMES:
Long-term Pain Control | Follow-up Visits up to 1-Year

CONTACTS AND LOCATIONS:
Overall Officials: Erik Kubiak, Principal Investigator — Orthopedic Surgery
Locations (1):
- University of Utah, Salt Lake City, Utah, United States